CLINICAL TRIAL: NCT05221671
Title: Impact of the Information Leaflet on the Preoperative Anesthesia Knowledge and Anxiety Levels of Children and Parents Before the Pediatric Endoscopic Procedures
Brief Title: Impact of the Information Leaflet on the Anesthesia Knowledge and Anxiety Levels of Children and Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Selin Erel, attending doctor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 184(13.12.2021)
Record Dates: First submitted 2021-12-23; First posted 2022-02-03 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2022-01

CONDITIONS: Anxiety; Preoperative Anxiety; Pediatric Anesthesia
Keywords: Anxiety; Anesthesia; Preoperative care; Child
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Patients and parents participating in the study will be divided into two groups by randomization. An information leaflets will be given to one group, but not to other group. Anesthesia knowledge level and anxiety level assessment questionnaires will be administered to both groups. These survey results will be compared between the two groups.
Who Masked: Investigator
Masking Description: The demographic data of the children and parents who agreed to participate in the study will be recorded by the anesthetist in the polyclinic, and an information leaflet will be given to those who will be included in the group that receives the information leaflet. Anesthesia knowledge level and anxiety level determination questionnaire and m-YPAS will be done by the researchers. Researchers applying these scales will not know which patients are included in the group receiving the information leaflet and which patients are in the control group. Conversion and evaluation of the survey results into study data will be done by other researchers. The principal researcher will supply the communication between these researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- not received information leaflet (No Intervention): During the preoperative anesthesia clinic examination, demographic data will be recorded and routine information about anesthesia will be provided. However, the information leaflet will not be handed to the patient and parents.
  The m-YPAS scale for pediatric patients will be evaluated and filled by the investigators before the anesthesia induction. Parents will be asked to fill out questionnaires for anxiety assessment and anesthesia knowledge level in the waiting room before the procedure.
- received information leaflet (Active Comparator): During the preoperative anesthesia evaluation, the children and their parents, who are included in the group who will receive information leaflets according to randomization, will be given information leaflets and both the child and their parents will be asked to read them before the procedure day. Age-appropriate brochures will be provided for children, and parent information leaflets will be provided for parents.
  The m-YPAS scale for pediatric patients will be evaluated and filled by the investigators before the anesthesia induction. Parents will be asked to fill out questionnaires for anxiety assessment and anesthesia knowledge level in the waiting room before the procedure.
  Interventions: Other: information leaflet

INTERVENTIONS:
Other: information leaflet — Leaflets prepared to inform about anesthesia and endoscopic procedure will be given to both parents and pediatric patients. A standard leaflet has been prepared for parents. Two leaflets have been prepared for children under the age of 12 and for adolescent patients over the age of 12. Unlike routine hospital information forms, all leaflets designed and prepared as a cartoon book. It is narrated using photographs of the materials and toys in the endoscopy room. It was predicted that there would be a difference between the groups who read and did not read this information leaflet in terms of anxiety levels and anesthesia knowledge levels.
  Arms: received information leaflet

SUMMARY:
The study includes applying a questionnaire to each child and their parents who applied to the anesthesia outpatient clinic for the gastroenterological endoscopic procedure. Children and parents will be divided into two groups, those who received and those who did not receive information leaflet. With the questionnaire both groups will be compared in terms of knowledge level and anxiety level.

DETAILED DESCRIPTION:
All children under the age of 18, who meet the inclusion criteria, applied to the outpatient clinic for the preoperative anesthesia evaluation will be included in the study. During the preoperative anesthesia examination, pediatric patients and their parents will be informed about the study, their consent will be obtained, and their demographic data will be recorded.

Information leaflets will be given to the one group in that both the child and their parents will read it before the endoscopic procedure. Children will handed leaflet appropriate for their age. The other group will not receive information leaflets. Routine information about anesthesia will be given to both groups.

Demographic data, m-YPAS(The modified Yale Preoperative Anxiety Scale), APAIS(Amsterdam Preoperative Anxiety and Information Scale) will be evaluated for both groups before anesthesia induction.

The anesthesiologist evaluate anxiety of children, will not know whether the patients received an information leaflets.

Parents will be asked to fill out the questionnaire in the waiting room. Anxiety scores will be evaluated by APAIS. The source of their knowledge about anesthesia, how anesthesia applications are made during endoscopy procedures and what their fears about anesthesia are will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All children under the age of 18 and their parents who applied to the anesthesia outpatient clinic before the gastroenterological endoscopic procedure
* Knowing Turkish language
* Agreeing to participate in the research voluntarily
* Parent and child not having a diagnosed neuropsychiatric disease
* Literacy of the child and parent
* Not having verbal communication barrier

Exclusion Criteria:

* Refusing to participate in the research
* Not knowing Turkish language
* Having a verbal communication barrier
* Parent and child have a diagnosed neuropsychiatric disease
* Illiteracy of the child or parent

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 142 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of preoperative anxiety scores of children with the Modified Yale Preoperative Anxiety Scale | Children's anxiety scale (m-YPAS) will be filled by the researcher observationally before the procedure.
  Leaflets have an effect on the anxiety score of children. Children who read information leaflet have lower anxiety scores than children who do not. Children's anxiety levels will be evaluated with the Modified Yale Preoperative Anxiety Scale (m-YPAS). This scale evaluates 22 items in 5 groups. The lowest score is 5, indicating the lowest level of anxiety. The highest score is 22, which indicates the most severe anxiety state.

SECONDARY OUTCOMES:
Evaluation of parents' knowledge and anxiety levels about anesthesia with the Amsterdam Preoperative Anxiety and Information Scale (APAIS) | Parents will be asked to fill out the anesthesia knowledge and anxiety level determination questionnaire in the waiting room before the endoscopy procedure.
  Anxiety levels are lower in children of parents who have higher level of knowledge and lower level of anxiety about anesthesia. The APAIS is a six-item questionnaire used to for the rapid assessment of preoperative anxiety. The APAIS consists of two scales that include a four-item anxiety scale and a two-item information requirement scale. The items are rated on a Likert scale from 1 ("not at all worrying") to 5 ("extremely worrying"). The score ranges of the anxiety subscale and information requirement subscale are 4-20 and 2-10, respectively. High scores are associated with high anxiety levels and information requirement.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University School of Medicine, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Overall results of research will be shared, individual answers of participants wont be shared.

REFERENCES:
- [Background] Kassai B, Rabilloud M, Dantony E, Grousson S, Revol O, Malik S, Ginhoux T, Touil N, Chassard D, Pereira de Souza Neto E. Introduction of a paediatric anaesthesia comic information leaflet reduced preoperative anxiety in children. Br J Anaesth. 2016 Jul;117(1):95-102. doi: 10.1093/bja/aew154. PMID 27317708
- [Background] Cumino Dde O, Cagno G, Goncalves VF, Wajman DS, Mathias LA. Impact of preanesthetic information on anxiety of parents and children. Braz J Anesthesiol. 2013 Nov-Dec;63(6):473-82. doi: 10.1016/j.bjane.2013.04.003. Epub 2013 Dec 5. PMID 24565345
- [Background] Landier M, Villemagne T, Le Touze A, Braik K, Meignan P, Cook AR, Morel B, Lardy H, Binet A. The position of a written document in preoperative information for pediatric surgery: A randomized controlled trial on parental anxiety, knowledge, and satisfaction. J Pediatr Surg. 2018 Mar;53(3):375-380. doi: 10.1016/j.jpedsurg.2017.04.009. Epub 2017 Apr 21. PMID 28456425